CLINICAL TRIAL: NCT01688362
Title: Platelet Rich Plasma vs. Corticosteroid Injection in the Treatment of Partial Thickness Rotator Cuff Tears. A Randomized, Prospective, Double Blinded Trial.
Brief Title: Platelet Rich Plasma vs. Corticosteroid Injection in the Treatment of Partial Rotator Cuff Tears
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Did not meet target enrollment deadlines.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-1016
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2016-02

CONDITIONS: Rotator Cuff Tear
Keywords: Prospective Randomized Controlled Double Blinded Trial; Rotator Cuff Tear; Platelet Rich Plasma; Corticosteroid; Ultrasound
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Adrenal Cortex Hormones; Bupivacaine; Triamcinolone Acetonide; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- platelet-rich plasma protein (PRP) (Experimental): Subjects in this group will receive 2 injections with PRP. Each injection separated by two weeks.
  Interventions: Biological: Platelet Rich Plasma (PRP)
- Corticosteroid (Active Comparator): Subjects in this group will receive one injection with corticosteroids and then one injection with local anesthetic two weeks later.
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Biological: Platelet Rich Plasma (PRP) — Subjects in this group will receive 2 injections with PRP. Subjects will have will have 15cc of blood drawn with the Arthrex ACP syringe. The blood will be placed into the Arthrex PRP centrifuge and spun at 1500 rpms for 5 minutes. The platelets will be drawn off to create the PRP for injection. A posterior glenohumeral injection under ultrasound guidance will be performed to inject the PRP solution using a 22g needle. A dry sterile dressing will be placed on the injection site. This injection will Take place at time zero and then two weeks later it will be repeated.
  Arms: platelet-rich plasma protein (PRP)
Drug: Corticosteroid — Subjects in this group will receive one injection with corticosteroids and then one injection with local anesthetic two weeks later. For the first injection patients will have 15ml of blood drawn. This blood will then be discarded in a biohazard container. A 6ml solution of 4ml 0.25% Bupivacaine, 1ml 40mg Kenalog, and 1ml 4mg Dexamethasone will be prepared. A posterior glenohumeral injection under ultrasound guidance will be performed to inject the steroid solution using a 22g needle. A dry sterile dressing will be placed at the injection site.
  For the second injection two weeks later patients will have 15 ml of blood drawn. This blood will then be discarded in a biohazard container. Using the same technique as in Visit 2, the investigator will inject a 6 ml solution of 2 ml sterile normal saline with 4 ml 0.25% Bupivacaine to the shoulder using ultrasound. A dry sterile dressing will be placed at the injection site.
  Other Names: Bupivacaine; Kenalog; Dexamethasone
  Arms: Corticosteroid

SUMMARY:
The purpose of this study is to further define the optimal non-surgical treatment strategy for partial thickness rotator cuff tears. The specific aim of this study is to determine the outcomes of treatment of partial thickness rotator cuff tears with corticosteroid or platelet rich plasma (PRP). Subjects with partial thickness rotator cuff tears will be randomized to receive an injection of PRP or corticosteroid. Shoulder function and tendon healing will be evaluated using the patient surveys as well as ultrasound. Subjects will be followed for one year to determine the outcomes for each treatment. The hypothesis is that there is no difference in healing rate or functional outcomes in patients treated with corticosteroid injections vs. PRP injections for the treatment of partial thickness rotator cuff tears.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain for at least two weeks.
* Partial thickness articular sided rotator cuff tear diagnosed by MRI and musculoskeletal ultrasound.

Exclusion Criteria:

* Prior surgery to the injured shoulder
* Full thickness rotator cuff tear
* Pregnancy
* Cancer
* Current treatment with anticoagulation medication
* Steroid injection in the past 6 months in the injured shoulder
* Prior PRP treatment to the injured shoulder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Percent change in Disabilities of the Arm, Shoulder, and Hand score. (DASH) | baseline and one year
  Disabilities of the Arm, Shoulder, and Hand (DASH) is a 30-item self-reported questionnaire used assess shoulder function. The DASH is widely used in orthopaedic research and is considered valid and reliable.

SECONDARY OUTCOMES:
Percent change in Disabilities of the Arm, Shoulder, and Hand score. (DASH) | baseline six weeks, 3 months, 6 months
Percent change in Visual Analog Pain scale (VAS) | Baseline, six weeks, three months, six months, one year
  Visual Analog Pain scale (VAS) is a self-reported questionnaire used to measure a patients pain level on a scale from 0 (no pain) to 10 (extreme pain).
Percent change in American Shoulder and Elbow Surgeons (ASES) scale | Baseline, six weeks, three months, six months, one year
  American Shoulder and Elbow Surgeons (ASES) scale is used to measure shoulder function. It is combines both physician assessment and patient self-reported questionnaire date to create the functional score.
Size of rotator cuff tear size. | Baseline, six months and one year
  Rotator cuff tear size will be determined using ultrasound imaging. The mean size at six months and one year will be compared to baseline per-treatment size.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan C Mackinnon-Patterson, BS, MPH, MD, Principal Investigator — University of North Carolina Department of Orthopaedics; Berkoff David, MD, Study Director — University of North Carolina Department of Orthopaedics
Locations (1):
- University of North Carolina Department of Orthopaedics, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Wolff AB, Sethi P, Sutton KM, Covey AS, Magit DP, Medvecky M. Partial-thickness rotator cuff tears. J Am Acad Orthop Surg. 2006 Dec;14(13):715-25. doi: 10.5435/00124635-200612000-00003. PMID 17148619
- [Background] Reilly P, Macleod I, Macfarlane R, Windley J, Emery RJ. Dead men and radiologists don't lie: a review of cadaveric and radiological studies of rotator cuff tear prevalence. Ann R Coll Surg Engl. 2006 Mar;88(2):116-21. doi: 10.1308/003588406X94968. PMID 16551396
- [Background] Sher JS, Uribe JW, Posada A, Murphy BJ, Zlatkin MB. Abnormal findings on magnetic resonance images of asymptomatic shoulders. J Bone Joint Surg Am. 1995 Jan;77(1):10-5. doi: 10.2106/00004623-199501000-00002. PMID 7822341
- [Background] Milgrom C, Schaffler M, Gilbert S, van Holsbeeck M. Rotator-cuff changes in asymptomatic adults. The effect of age, hand dominance and gender. J Bone Joint Surg Br. 1995 Mar;77(2):296-8. PMID 7706351
- [Background] Teefey SA, Rubin DA, Middleton WD, Hildebolt CF, Leibold RA, Yamaguchi K. Detection and quantification of rotator cuff tears. Comparison of ultrasonographic, magnetic resonance imaging, and arthroscopic findings in seventy-one consecutive cases. J Bone Joint Surg Am. 2004 Apr;86(4):708-16. PMID 15069134
- [Background] Sheth U, Simunovic N, Klein G, Fu F, Einhorn TA, Schemitsch E, Ayeni OR, Bhandari M. Efficacy of autologous platelet-rich plasma use for orthopaedic indications: a meta-analysis. J Bone Joint Surg Am. 2012 Feb 15;94(4):298-307. doi: 10.2106/JBJS.K.00154. PMID 22241606
- [Background] GlobalData. Platelet rich plasma: a market snapshot. http://www.docstoc.com/docs/47503668/Platelet-Rich-Plasma-A-Market-Snapshot. September 12, 2012.
- [Background] Jo CH, Kim JE, Yoon KS, Shin S. Platelet-rich plasma stimulates cell proliferation and enhances matrix gene expression and synthesis in tenocytes from human rotator cuff tendons with degenerative tears. Am J Sports Med. 2012 May;40(5):1035-45. doi: 10.1177/0363546512437525. Epub 2012 Feb 23. PMID 22366517
- [Background] Chahal J, Van Thiel GS, Mall N, Heard W, Bach BR, Cole BJ, Nicholson GP, Verma NN, Whelan DB, Romeo AA. The role of platelet-rich plasma in arthroscopic rotator cuff repair: a systematic review with quantitative synthesis. Arthroscopy. 2012 Nov;28(11):1718-27. doi: 10.1016/j.arthro.2012.03.007. Epub 2012 Jun 12. PMID 22694941
- [Background] Randelli P, Arrigoni P, Ragone V, Aliprandi A, Cabitza P. Platelet rich plasma in arthroscopic rotator cuff repair: a prospective RCT study, 2-year follow-up. J Shoulder Elbow Surg. 2011 Jun;20(4):518-28. doi: 10.1016/j.jse.2011.02.008. PMID 21570659
- [Background] Castricini R, Longo UG, De Benedetto M, Panfoli N, Pirani P, Zini R, Maffulli N, Denaro V. Platelet-rich plasma augmentation for arthroscopic rotator cuff repair: a randomized controlled trial. Am J Sports Med. 2011 Feb;39(2):258-65. doi: 10.1177/0363546510390780. Epub 2010 Dec 15. PMID 21160018
- [Background] Peerbooms JC, Sluimer J, Bruijn DJ, Gosens T. Positive effect of an autologous platelet concentrate in lateral epicondylitis in a double-blind randomized controlled trial: platelet-rich plasma versus corticosteroid injection with a 1-year follow-up. Am J Sports Med. 2010 Feb;38(2):255-62. doi: 10.1177/0363546509355445. PMID 20448192
- [Background] Gosens T, Peerbooms JC, van Laar W, den Oudsten BL. Ongoing positive effect of platelet-rich plasma versus corticosteroid injection in lateral epicondylitis: a double-blind randomized controlled trial with 2-year follow-up. Am J Sports Med. 2011 Jun;39(6):1200-8. doi: 10.1177/0363546510397173. Epub 2011 Mar 21. PMID 21422467
- [Background] Wolf JM, Ozer K, Scott F, Gordon MJ, Williams AE. Comparison of autologous blood, corticosteroid, and saline injection in the treatment of lateral epicondylitis: a prospective, randomized, controlled multicenter study. J Hand Surg Am. 2011 Aug;36(8):1269-72. doi: 10.1016/j.jhsa.2011.05.014. Epub 2011 Jun 25. PMID 21705157
- [Background] de Vos RJ, Weir A, van Schie HT, Bierma-Zeinstra SM, Verhaar JA, Weinans H, Tol JL. Platelet-rich plasma injection for chronic Achilles tendinopathy: a randomized controlled trial. JAMA. 2010 Jan 13;303(2):144-9. doi: 10.1001/jama.2009.1986. PMID 20068208
- [Background] de Jonge S, de Vos RJ, Weir A, van Schie HT, Bierma-Zeinstra SM, Verhaar JA, Weinans H, Tol JL. One-year follow-up of platelet-rich plasma treatment in chronic Achilles tendinopathy: a double-blind randomized placebo-controlled trial. Am J Sports Med. 2011 Aug;39(8):1623-9. doi: 10.1177/0363546511404877. Epub 2011 May 21. PMID 21602565
- [Background] Alvarez CM, Litchfield R, Jackowski D, Griffin S, Kirkley A. A prospective, double-blind, randomized clinical trial comparing subacromial injection of betamethasone and xylocaine to xylocaine alone in chronic rotator cuff tendinosis. Am J Sports Med. 2005 Feb;33(2):255-62. doi: 10.1177/0363546504267345. PMID 15701612